CLINICAL TRIAL: NCT01714596
Title: A Prospective Randomized Trial to Assess PO Versus IV Antibiotics for the Treatment of Post-op Wound Infection After Extremity Fractures (POvIV)
Brief Title: Randomized Trial to Assess PO Versus IV Antibiotics
Acronym: POvIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Major Extremity Trauma Research Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: METRC POvIV
Record Dates: First submitted 2012-04-30; First posted 2012-10-26 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Wound Infection
Keywords: Oral Antibiotic; Intravenous Antibiotic; Wound infection; Randomized Controlled Trial
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral Antibiotic (Active Comparator): Oral Antibiotic Arm; Participants assigned to this group will receive oral antibiotics as prescribed by their treating physician.
  Interventions: Other: PO versus IV antibiotics Route of administration evaluation
- IV Antibiotic (Active Comparator): Participants assigned to this group will receive intravenous (IV) antibiotics as prescribed by their treating physician.
  Interventions: Other: PO versus IV antibiotics Route of administration evaluation

INTERVENTIONS:
Other: PO versus IV antibiotics Route of administration evaluation — This is a study of oral (per os, (PO)) antibiotic therapy versus intravenous (IV) antibiotics in the treatment of acute infection after fixation of fractures and joint fusions. This is not a study of an experimental drug but a study of route of administration of standard use antibiotics. Antibiotic regimen options decision will be made by the Study Surgeon at each site in consult with local Infectious Disease experts based on local standard practices and bacterial susceptibilities.
  Other Names: based on local practices and bacterial susceptibilities

SUMMARY:
The goal of this study is to evaluate the effect of treatment of post-op wound infection in long bones after fracture fixation or joint fusion and either: (Group 1) operative debridement and PO antibiotic treatment for 6 weeks; or (Group 2) operative debridement and IV antibiotics for 6 weeks.

Primary Hypothesis 1: The rate of study injury related surgical interventions by one year in Group 1 will be non-inferior to the rate in Group 2.

Secondary Hypothesis 1: The rate of treatment failure by one year in Group 1 will be non-inferior to the rate in Group 2. Treatment failure is defined as wound problems that require surgery >2 weeks after initial debridement, infection recurrence, infection with a new pathogen, joint erosion, implant failure, medical problems related to the treatment administration which necessitates a switch from one arm to the other.

Secondary Hypothesis 2: The rate of re-hospitalization for complications, infection, non-union and amputation by one year in Group 1 will be non-inferior to the rate in Group 2.

Secondary Hypothesis 3: Following discharge for treatment of infection, per patient treatment costs at 1 year will be lower in Group 1 than in Group 2.

Secondary Hypothesis 4: Adherence in Group 1 will be non-inferior to adherence in Group 2.

Secondary Hypothesis 5: Patient satisfaction with treatment in Group 1 will be non-inferior to adherence in Group 2.

Specific Aim 2: To build and validate a risk prediction model for failure of treatment of early post-op wound infections after fixation of fractures and joint fusions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with any fractures of any bone at or proximal to and including the tarsal/metatarsal joint (Lisfranc) or proximal to the carpal joints (includes distal radius fractures), excluding the spine, treated with any type of internal fixation, or
2. Patients undergoing fusion of any bone at or proximal to and including the subtalar joint or radial carpal joint, (excluding the spine) that develop a post op wound infection at any time.
3. Patients diagnosed with a wound infection of the study injury, defined as patients with at least one of the following:

   1. Deep culture positive after operative debridement.
   2. Cultures positive in thio only after operative debridement.
   3. Negative culture after operative debridement if wound infection meets the Center for Disease control and Prevention (CDC) criteria.
4. Patients who are English or Spanish competent.
5. Patients aged 18 - 84.
6. Patients with bacteria susceptible to both PO and IV antibiotics.
7. Patients able to be treated for their infection at the METRC facility for at least 12 months following definitive surgical procedure
8. Patients may have multiple eligible study-eligible injuries.
9. Patients may have temporary external fixation prior to definitive fixation.
10. Patients may have received antibiotics prior to operative wound debridement.
11. Patient is able to obtain study medication(s).
12. Patient may be pregnant at the time of screening.

Exclusion Criteria:

1. Patients who have high risk of amputation of the study limb (based on opinion of the initial managing physician).
2. Patients undergoing treatment with any other investigational therapy within the month preceding implantation or planned within the 12 months following implantation.
3. Patients with history of chronic infection at the site of study injury, defined as:

   patients with chronic osteomyelitis identified by radiographic erosion or sequestrum; or patients with more than one instance of surgical treatment of infection and approximately 6 week course of antibiotics.
4. Patients with pathological fractures; a known history of Paget's disease.
5. Patients for whom the definitive treatment of the study injury was an external fixator.
6. Patients who are currently on Selective Serotonin Reuptake Inhibitor (SSRI) medication (e.g. Zoloft, Prozac, Celexa), and bacteria is MRSA
7. Patients with cultures positive in thio only.
8. Patients who are incarcerated or who have unstable housing situations due to concerns regarding ability to receive home care, adherence phone calls, and maintain follow up. .
9. Patients or designated proxy who are unwilling to provide consent.
10. Patients with a history of IV drug use who in the investigator's opinion are unsuitable candidates for IV therapy.
11. Patients likely to have severe problems maintaining follow-up, including patients diagnosed with a severe psychiatric conditions, patients who live too far outside the hospital's catchment area.
12. Patients with traumatic brain injury or who are intellectually challenged and who lack adequate family support to ensure adherence to the protocol.
13. Patients unable to swallow oral medications or without adequately functioning GI tract.
14. Patients who, based upon the clinical judgment of the treating clinician, are NOT equally suited for treatment with either oral or intravenous antibiotics (i.e., those for whom there is a clinical treatment preference).

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2013-12-03 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Study injury related surgical interventions by 1 year | 1 year

SECONDARY OUTCOMES:
Treatment Failure by 1 year | 1 year
  Treatment failure is defined as wound problems that require surgery >2 weeks after initial debridement, infection recurrence, infection with a new pathogen, joint erosion, implant failure, medical problems related to the treatment administration which necessitates a switch from one arm to the other.
Re-hospitalizations by 1 year | 1 year
  Re-hospitalization for complications, such as infection, non-union and amputation
Healthcare costs | 1 year
  Cost of PO versus IV medications include medical record and bill abstracted costs associated with outpatient clinic visits, home health visits, medication, subsequent hospital readmission, and other types of medical care as identified over the course of the study.
Medication Adherence | 1 year
  Patient adherence to PO and IV medications
  Patient adherence with PO antibiotics will be monitored through wireless-enabled microchip monitors embedded in pill bottles by the Medication Event Monitoring System (MEMS) and weekly adherence questionnaire.
Satisfaction with treatment | 1 year
  Patient satisfaction with treatment measured by Short Form Patient Satisfaction Questionnaire (PSQ-18)
  The PSQ-18 measures 6 domains: technical quality, interpersonal manner, communication, financial aspects of care, time spent with doctor, and accessibility. A score of 0.8 or higher in each domain correlates with improved satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: William T Obremskey, MD, Principal Investigator — Vanderbilt University Medical Center; Renan Castillo, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Tara Taylor, MPH, Study Director — Johns Hopkins Bloomberg School of Public Health
Locations (24):
- United States (24):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - Denver Health and Hospital Authority, Denver, Colorado
  - University of Miami Ryder Trauma Center, Miami, Florida
  - Eskenazi Health, Indianapolis, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Maryland R Adams Cowley Shock Trauma Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - St. Louis University Medical Center, St Louis, Missouri
  - Jamaica Hospital Medical Center, Jamaica, New York
  - NYU Langone Medical Center, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Penn State University M.S. Hershey Medical Center, Hershey, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - San Antonio Military Medical Center (SAMMC), San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Naval Medical Center Portsmouth, Portsmouth, Virginia
  - University of Washington/Harborview Medical Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Derived] Major Extremity Trauma Research Consortium (METRC); Obremskey WT, O'Toole RV, Morshed S, Tornetta P 3rd, Murray CK, Jones CB, Scharfstein DO, Taylor TJ, Carlini AR, DeSanto JM, Castillo RC, Bosse MJ, Karunakar MA, Seymour RB, Sims SH, Weinrib DA, Churchill C, Carroll EA, Pilson HT, Goodman JB, Holden MB, Miller AN, Sietsema DL, Stahel PF, Mir H, Schmidt AH, Westberg JR, Mullis B, Shively KD, Hymes RA, Konda SR, Vallier HA, Breslin MA, Smith CS, Crickard CV, Reid JS, Baker M, Eglseder WA, LeBrun C, Manson T, Mascarenhas DC, Nascone J, Pollak AN, Schloss MG, Sciadini MF, Degani Y, Miclau T, Weiss DB, Yarboro SR, McVey ED, Firoozabadi R, Agel J, Burgos EJ, Gajari V, Rodriguez-Buitrago A, Tummuru RR, Trochez KM. Oral vs Intravenous Antibiotics for Fracture-Related Infections: The POvIV Randomized Clinical Trial. JAMA Surg. 2025 Mar 1;160(3):276-284. doi: 10.1001/jamasurg.2024.6439. PMID 39841468